CLINICAL TRIAL: NCT04759989
Title: Fluid Resuscitation in Septic Shock Patients With BMI Elevation
Acronym: FRISSBE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is being closed due to low enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fluid resuscitation
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Sepsis; Septic Shock; Obesity
MeSH Terms: conditions — Sepsis; Shock, Septic; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30cc/kg ideal body weight (IBW) (Active Comparator): 30cc/kg intravenous fluids based on the patients calculated ideal body weight will be administered when randomized to this arm
  Using Devine's formula. (men: 50kg + 2.3kg * (height(in) - 60); women: 45.5kg + 2.3kg * (height(in) - 60)
  Interventions: Procedure: Ideal Body Weight Dosing
- 30cc/kg adjusted body weight (AdjBW) (Active Comparator): 30cc/kg intravenous fluids based on the patients calculated adjusted body weight will be administered when randomized to this arm
  Calculated by the following formula: AdjBW = IBW + 0.4(ABW - IBW).
  Interventions: Procedure: Adjusted Body Weight Dosing
- 30cc/kg actual body weight (ABW) (Active Comparator): 30cc/kg intravenous fluids based on the patients actual body weight will be administered when randomized to this arm
  Patients will receive an initial fluid bolus of 30 cc/kg of actual body weight
  Interventions: Procedure: Actual Body Weight Dosing

INTERVENTIONS:
Procedure: Actual Body Weight Dosing — 30cc/kg initial bolus calculated using Actual Body Weight
  Arms: 30cc/kg actual body weight (ABW)
Procedure: Adjusted Body Weight Dosing — 30cc/kg initial bolus calculated using Adjusted Body Weight
  Arms: 30cc/kg adjusted body weight (AdjBW)
Procedure: Ideal Body Weight Dosing — 30cc/kg initial bolus calculated using Ideal Body Weight
  Arms: 30cc/kg ideal body weight (IBW)

SUMMARY:
To explore the safety and feasibility of alternative fluid resuscitation strategies in obese patients with septic shock.

DETAILED DESCRIPTION:
Early, goal-directed therapy with timely achievement of hemodynamic stability has been shown to clearly improve outcomes in patients with septic shock. Although Surviving Sepsis Campaign guidelines recommend a weight-based approach to initial fluid resuscitation (i.e. 30ml/kg),1 at present, there are no robust data to support whether dosing based on actual body weight or an alternative correction formula (ideal body weight, adjusted body weight) is superior.

FRISSBE is a prospective, randomized, three-arm parallel-group pilot trial of alternative resuscitation strategies for obese patients with septic shock, looking at feasibility and safety of different weight-based approaches. Subject treatment assignment will not be blinded. Data will be collected and analyzed on an intent-to-treat basis. The study will enroll 60 subjects, with 20 subjects per treatment arm. Subjects will be randomized to receive one of three weight-based initial fluid resuscitation strategies - 30cc/kg ideal body weight (IBW), 30cc/kg adjusted body weight (AdjBW), or 30cc/kg actual body weight (ABW).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* BMI > 30
* suspected infection, and either:

  * hypotension (a systolic blood pressure < 90mmHg) or
  * blood lactate concentration > 4mmol/L

Exclusion Criteria:

* Pregnant
* Primary diagnosis of acute cerebral vascular event
* Acute coronary syndrome
* Acute pulmonary edema
* Status asthmaticus
* Major cardiac arrhythmia
* Active gastrointestinal hemorrhage
* Seizures
* Drug overdose
* Burns or trauma
* Requirement for immediate surgery
* CD4<50/mm3
* Do-not-resuscitate order status
* Transferred from another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Feasibility1: fluid target | 3 hours
  percentage of of patients with actual volume received within 10% of target fluid volume.
Safety-ventilation | 24 hours
  Proportion of patients requiring invasive or noninvasive mechanical ventilation
Safety-vasopressors | 24 hours
  proportion of patients requiring vasopressor administration
Safety-time to hemodynamic stability | 72 hours
  time from randomization to map >65 without use of vasopressors and no lactate >2

SECONDARY OUTCOMES:
Exploratory: in-hospital all cause mortality | 28 days
  Proportion of patient in each group who experience death due to any cause during hospitalization up to 28 days
Exploratory: ICU length of stay | 28 days
  number of consecutive midnights in ICU
feasibility2: recruitment rate | study duration
  proportion of patients enrolled out of patients screened to randomized through completion of study, an average of 1 year
feasibility3: time to randomization | 3 hours
  median time from screening to randomization
Exploratory: hospital length of stay | 28 days
  number of midnights spent in hospital up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Brice Taylor, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Background] Wacharasint P, Boyd JH, Russell JA, Walley KR. One size does not fit all in severe infection: obesity alters outcome, susceptibility, treatment, and inflammatory response. Crit Care. 2013 Jun 20;17(3):R122. doi: 10.1186/cc12794. PMID 23786836
- [Background] Arabi YM, Dara SI, Tamim HM, Rishu AH, Bouchama A, Khedr MK, Feinstein D, Parrillo JE, Wood KE, Keenan SP, Zanotti S, Martinka G, Kumar A, Kumar A; Cooperative Antimicrobial Therapy of Septic Shock (CATSS) Database Research Group. Clinical characteristics, sepsis interventions and outcomes in the obese patients with septic shock: an international multicenter cohort study. Crit Care. 2013 Apr 17;17(2):R72. doi: 10.1186/cc12680. PMID 23594407
- [Background] Boyd JH, Forbes J, Nakada TA, Walley KR, Russell JA. Fluid resuscitation in septic shock: a positive fluid balance and elevated central venous pressure are associated with increased mortality. Crit Care Med. 2011 Feb;39(2):259-65. doi: 10.1097/CCM.0b013e3181feeb15. PMID 20975548
- [Background] Marik PE, Linde-Zwirble WT, Bittner EA, Sahatjian J, Hansell D. Fluid administration in severe sepsis and septic shock, patterns and outcomes: an analysis of a large national database. Intensive Care Med. 2017 May;43(5):625-632. doi: 10.1007/s00134-016-4675-y. Epub 2017 Jan 27. PMID 28130687
- [Background] Taylor SP, Karvetski CH, Templin MA, Heffner AC, Taylor BT. Initial fluid resuscitation following adjusted body weight dosing is associated with improved mortality in obese patients with suspected septic shock. J Crit Care. 2018 Feb;43:7-12. doi: 10.1016/j.jcrc.2017.08.025. Epub 2017 Aug 15. PMID 28823951